CLINICAL TRIAL: NCT01232036
Title: A Clinical Trial to Compare the Pharmacokinetic and Pharmacodynamic Characteristics and Safety After Oral Administration of Glucophage With Those After Oral Administration of HL-018 in Healthy Male Volunteers
Brief Title: Clinical Trial to Compare the Pharmacokinetics and Pharmacodynamics After Oral Administration of Glucophage and HL-018
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Medical Affairs Department, HanAll Biopharma Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-0195
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Reference
  Interventions: Drug: Glucophage 500mg
- B (Experimental): Test
  Interventions: Drug: HL-018 500mg
- C (Placebo Comparator): Placebo
  Interventions: Other: No administration of Drug

INTERVENTIONS:
Drug: Glucophage 500mg — Single Oral Dose of
  Arms: A
Drug: HL-018 500mg — Single Oral Dose of
  Arms: B
Other: No administration of Drug
  Arms: C

SUMMARY:
This study is designed to to compare the pharmacokinetic and pharmacodynamic characteristics and safety after oral administration of Glucophage with those after oral administration of HL-018 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 19 to 50 years at screening.
* No significant congenital/chronic disease. No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
* History of known hypersensitivity to drugs including metformin.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUClast and Cmax) | 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr